CLINICAL TRIAL: NCT03290274
Title: Clinical Trial to Evaluate the Efficacy and Security of Deep Brain Stimulation in Alzheimer´s Disease
Acronym: ECP-EA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital San Carlos, Madrid (Other)
Responsible Party: Principal Investigator, Juan Antonio Barcia Albacar, Head of Neurosurgery Department, Hospital San Carlos, Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ECP-EA
Record Dates: First submitted 2017-09-13; First posted 2017-09-21 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2017-08

CONDITIONS: Alzheimer Disease
Keywords: Deep brain stimulation; Alzheimer´s Disease; Fornix; Basal nucleus of Meynert
MeSH Terms: conditions — Alzheimer Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep brain stimulation (fornix) (Experimental): Deep brain stimulation at fornix area
  Interventions: Device: Deep brain stimulation (fornix)
- Deep brain stimulation (Basal nucleus of Meynert) (Experimental): Deep brain stimulation at Basal nucleus of Meynert
  Interventions: Device: Deep brain stimulation (Basal nucleus of Meynert)

INTERVENTIONS:
Device: Deep brain stimulation (fornix) — Deep brain stimulation at fornix
  Arms: Deep brain stimulation (fornix)
Device: Deep brain stimulation (Basal nucleus of Meynert) — Deep brain stimulation AT Basal nucleus of Meynert
  Arms: Deep brain stimulation (Basal nucleus of Meynert)

SUMMARY:
Approximately one million of Spaniards suffer from AlzhEimer´s Disease (AD) and this figure is expected to triple by 20150. The approved treatments modulate neurotransmission in general and are not specific or anatomically directed. In AD there is a dysfunction in cognitive and memory circuits. It has been shown that the deep brain stimulation (DBS) can specially modulate circuits in such a way that is modulable, and this approach is safe. The safety of this treatment and its biological effects are convincing enough to require further study of possible therapeutic effects of DBS in AD. The objectives are: To evaluate the security of DBS in AD (main objective). To study the influence of DBS in the progress of AD, to compare the effects of DBS on the brain metabolism neural connectivity and hubs using MEG, and to compare the effects between two different groups: fornix and Basal nucleus of Meynert (BNM). To achieve this, a prospective, double-blind comparison study between groups will be conducted, to evaluate the effects of DBS in 6 patients: group I (fornix) and group II ( BNM).

ELIGIBILITY:
Inclusion Criteria:

* Age: Between 50-80 years old
* Diagnosis criteria of Alzheimer disease (Dubois criteria) in the previous 2 years
* Presence of tau, p-tau or Aβ in cerebrospinal fluid or positive amiloid-PET scan
* Clinical dementia rating scale (CDR): 1
* Use of cholinesterase inhibitors and/or memantine during one year at least, and worsening in neuropsychologic tests in spite of the treatment
* Informed consent (patient and caregiver or legal representative)

Exclusion Criteria:

* Brain structural disorders: primary or metastatic tumor, Hydrocephalus, stroke, brain abscess or cerebral malformation
* Vascular dementia (NINCDS-AIREN criteria)
* Neurodegenerative disease other than AD
* Psychiatric disease
* Epilepsy
* Severe or unstable comorbidity (mellitus diabetes, high blood pressure…)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Security | 2 years
  Determinate number of adverse event in each group such as infections, hospitalization, epilepsia, bleeding or hemiparesis

CONTACTS AND LOCATIONS:
Overall Officials: Aurora Viloria, MD, Principal Investigator — Hospital Clinico San Carlos
Locations (1):
- Hospital Clinico San Carlos, Madrid, Spain

REFERENCES:
- [Derived] Barcia JA, Viloria MA, Yubero R, Sanchez-Sanchez-Rojas L, Lopez A, Strange BA, Cabrera M, Canuet L, Gil P, Nombela C. Directional DBS of the Fornix in Alzheimer's Disease Achieves Long-Term Benefits: A Case Report. Front Aging Neurosci. 2022 Apr 1;14:809972. doi: 10.3389/fnagi.2022.809972. eCollection 2022. PMID 35431895